CLINICAL TRIAL: NCT00807014
Title: Single-blind, Multicenter, Parallel, Comparative, Randomized, Phase 4 Clinical Trial for the Evaluation of the Quality of Life, Efficacy and Tolerance of Duac® Gel Against Differin® Gel in the Topical Treatment of Mild to Moderate Acne Vulgaris.
Brief Title: Evaluation of Quality of Life, Efficacy, and Tolerance of Duac® Gel Compared to Differin® Gel in the Treatment of Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114567; S194-SP-05/Duac
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: Differin; quality of life; Acne; Duac; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination; Adapalene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duac Gel (Experimental): Duac Gel
  Interventions: Drug: Duac Gel
- Differin gel (Active Comparator): Differin gel
  Interventions: Drug: Differin gel

INTERVENTIONS:
Drug: Duac Gel — Duac® Gel will be applied to the face once daily at night, for 12 weeks.
  Other Names: Duac
  Arms: Duac Gel
Drug: Differin gel — Differin Gel will be applied to the face once daily at night, for 12 weeks.
  Other Names: Differin
  Arms: Differin gel

SUMMARY:
The objectives of this clinical trial are to compare the quality of life of the subjects, the efficacy and the tolerance of Duac® Gel (gel formulation with a combination of clindamycin phosphate [equivalent to 1% clindamycin] and 5% benzoyl peroxide), applied once daily, against Differin® Gel (gel with 0.1% adapalene), used once daily, in the treatment of mild to moderate acne vulgaris.

DETAILED DESCRIPTION:
Acne vulgaris is a chronic inflammatory disease of the pilosebaceous unit. It is characterized by the formation of comedones, papules, pustules, nodules, cysts, maculae and scars, generally located on the face, chest and back. Acne pathogenesis is recognized as multifactorial.

Acne vulgaris is the most common dermatological disorder. It affects approximately 85% individuals at some point in their lives, generally between 12 and 24 years of age. Although acne is prevalent within this age range, it can persist for many years and its long-term physical and psychological implications can be significant.

There are several medicinal products used to treat acne. However, the therapeutic challenge remains, therefore it is essential to continue investigating effective strategies for the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild to moderate acne vulgaris on the face,.
* Subjects of either sex aged between 12 and 39 years, inclusive.
* Subjects agreeing not to use sun-beds or undergo any UV light treatment for 4 weeks prior to entering the study and to minimize the amount of exposure to direct sunlight for the duration of the study.

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or sexually active with the potential to have children, and not using a contraception method that is safe from a medical point of view
* Subjects using anti-androgen containing contraceptives.
* Subjects who, during the past month, have received oral or topical steroids or antibiotics, or acne treatment of any type, including natural or artificial UV therapy.
* Subjects who have a history of hypersensitivity or idiosyncratic reaction to clindamycin phosphate, benzoyl peroxide, adapalene or any components of the medicinal products which will be used during the study.
* Subjects using, or having used in the past month, any significant concomitant medicinal product which might affect their acne, as judged by the Investigator.
* Subjects with a history of regional enteritis or ulcerative colitis, or a history of antibiotic-associated colitis.
* Subjects with a history of photosensitivity.

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 169 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Spain (8):
  - Hospital Abente y Lago in La Coruna, A Coruña
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Ramón and Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario Ntra. Sra. de the Victoria, Málaga
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Clínico de Salamanca, Salamanca

RESULTS

PARTICIPANT FLOW:
Groups:
- Duac Gel: Duac gel (combination of clindamycin phosphate [equivalent to 1% clindamycin] and 5% benzoyl peroxide) applied topically to facial acne once nightly for 12 weeks
- Differin Gel: Differin gel (containing 0.1% adapalene) applied topically to facial acne once nightly for 12 weeks
Period: Overall Study
Arm/Group | Duac Gel | Differin Gel
Started | 83 | 85
Completed | 56 | 58
Not Completed | 27 | 27
Not completed — Participant Considered Disease Cured | 13 | 2
Not completed — Participant Considered Disease Not Cured | 2 | 7
Not completed — Protocol Violation | 2 | 8
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 9 | 7
Not completed — Recovery | 1 | 0
Not completed — Missed Visit 2 Due to Personal Reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duac Gel | Differin Gel | Total
Number analyzed (Participants) | 83 | 85 | 168
Age Continuous [Mean (Standard Deviation); unit: Years] | 18.9 (5.3) | 19.2 (5.3) | 19.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 65 | 124
  Male | 24 | 20 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 75 | 77 | 152
  Asian | 2 | 1 | 3
  Black | 1 | 0 | 1
  Mixed or Multiracial | 2 | 3 | 5
  Captured as "Other" on Case Report Form | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 2 in the Global Score of the Participant-completed Skindex-29 Quality of Life (QoL) Questionnaire
Description: Skindex-29 is a self-administered QoL questionnaire comprised of 29 items scored on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=all the time) covering 3 domains: emotional (10 items), symptomatic (7 items), and functional (12 items), with domain scores ranging from 0 to 40, 28, and 48, respectively. Lower scores = better QoL. A Global Score (range 0-100) was derived by multiplying the sum of the points for all 29 items by a constant (0.862). Change from Baseline was calculated as the value at Week 2 minus the value at Baseline (Week 0).
Time Frame: Baseline (Week 0) and Week 2
Population: Intent-to-Treat (ITT) Population: all randomized participants (par.) who applied >= 1 dose of study product. Missing values were imputed using the last observation carried forward (LOCF, i.e., the last available observation was used to estimate subsequent missing data points) method. 1 par. in the Differin arm had no QoL data and was not analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 84
scores on a scale | -4.9 (7.2) | -1.1 (8.4)
Statistical Analysis 1: Comparison: Duac Gel vs Differin Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Analysis of covariance (ANCOVA) model was used with terms for baseline value, treatment, and center. Treatment-by-center interaction was not included

2. Secondary Outcome: Mean Change From Baseline to Week 12 for the Indicated Domain Scores and the Global Score of the Participant-completed Skindex-29 QoL Questionnaire
Description: as for outcome 1
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population. Missing values were imputed using the LOCF method (i.e., the last available observation was used to estimate subsequent missing data points). One participant in the Differin arm had no QoL data available and was thus excluded from analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 84
scores on a scale
  Symptomatic Domain | -7.4 (13.0) | -2.8 (16.7)
  Emotional Domain | -10.3 (15.1) | -5.4 (13.5)
  Functional Domain | -3.5 (7.6) | -0.1 (8.0)
  Global Score | -6.8 (9.1) | -2.6 (9.8)

3. Secondary Outcome: Mean Change From Baseline to Weeks 1, 2, 4, 8, and 12 in Inflammatory, Non-inflammatory, and Total Lesion Counts
Description: Lesions were counted on the entire face (defined as the area from the upper part of the jaw to the lower part of the hairline), excluding maculae and non-inflammatory lesions located on the nose or chin. Inflammatory lesions included papules, pustules, nodules, and cysts. Non-inflammatory lesions included closed comedones (whiteheads) and open comedones (blackheads). The total lesion count was calculated as the sum of inflammatory and non-inflammatory lesions. Change from Baseline was calculated as the values at Weeks 1, 2, 4, 8, and 12 minus the value at Baseline (Week 0).
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 8, and 12
Population: ITT Population. Missing values were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 85
lesions
  Non-inflammatory Lesions, Week 1 | -8.5 (12.8) | -6.3 (15.6)
  Non-inflammatory Lesions, Week 2 | -11.8 (17.3) | -8.2 (17.9)
  Non-inflammatory Lesions, Week 4 | -16.3 (20.2) | -9.1 (16.8)
  Non-inflammatory Lesions, Week 8 | -18.4 (21.7) | -8.4 (30.7)
  Non-inflammatory Lesions, Week 12 | -22.6 (23.0) | -12.6 (33.3)
  Inflammatory Lesions, Week 1 | -10.1 (12.5) | -5.4 (8.9)
  Inflammatory Lesions, Week 2 | -13.0 (13.2) | -8.5 (11.1)
  Inflammatory Lesions, Week 4 | -16.6 (14.4) | -9.6 (11.7)
  Inflammatory Lesions, Week 8 | -17.5 (16.1) | -8.7 (14.4)
  Inflammatory Lesions, Week 12 | -18.8 (17.8) | -11.2 (15.5)
  Total Lesions, Week 1 | -18.6 (18.1) | -11.7 (19.1)
  Total Lesions, Week 2 | -24.8 (21.0) | -16.8 (23.7)
  Total Lesions, Week 4 | -32.9 (25.2) | -18.8 (21.1)
  Total Lesions, Week 8 | -35.9 (29.0) | -17.1 (36.8)
  Total Lesions, Week 12 | -41.4 (32.3) | -23.8 (40.5)

4. Secondary Outcome: Mean Percent Change From Baseline to Weeks 1, 2, 4, 8, and 12 in Inflammatory, Non-inflammatory, and Total Lesion Counts
Description: Lesions were counted on the entire face (defined as the area from the upper part of the jaw to the lower part of the hairline), excluding maculae and non-inflammatory lesions located on the nose or chin. Inflammatory lesions (IL) included papules, pustules, nodules, and cysts. Non-inflammatory lesions (NIL) included closed comedones (whiteheads) and open comedones (blackheads). Total lesion count was calculated as the sum of IL and NIL. Percent change from Baseline was calculated as the values at Weeks 1, 2, 4, 8, and 12 minus the value at Baseline divided by Baseline value * 100.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 8, and 12
Population: ITT Population. Missing values were imputed using the LOCF method. Some participants had no baseline lesions of an individual type; percent change from baseline is undefined for these participants. All participants, however, had at least one type of lesion; thus, all participants in the ITT Population were analyzed for total lesion count.
Measure: Mean (Standard Deviation); unit: percent change in lesions
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 85
percent change in lesions
  Non-inflammatory Lesions, Week 1, n=74, 73 | -29.8 (36.3) | -22.9 (52.8)
  Non-inflammatory Lesions, Week 2, n=74, 73 | -38.4 (60.1) | -26.5 (79.5)
  Non-inflammatory Lesions, Week 4, n=74, 73 | -52.6 (50.7) | -36.4 (62.1)
  Non-inflammatory Lesions, Week 8, n=74, 73 | -59.5 (44.1) | -32.8 (68.9)
  Non-inflammatory Lesions, Week 12, n=74, 73 | -69.7 (36.4) | -45.5 (69.3)
  Inflammatory Lesions, Week 1, n=82, 84 | -36.8 (32.1) | -21.0 (45.1)
  Inflammatory Lesions, Week 2, n=82, 84 | -53.0 (32.7) | -36.4 (48.2)
  Inflammatory Lesions, Week 4, n=82, 84 | -67.9 (27.7) | -38.3 (50.6)
  Inflammatory Lesions, Week 8, n=82, 84 | -67.6 (31.4) | -33.8 (61.2)
  Inflammatory Lesions, Week 12, n=82, 84 | -72.4 (34.7) | -46.5 (58.5)
  Total Lesions, Week 1, n=83, 85 | -32.1 (28.6) | -22.6 (34.8)
  Total Lesions, Week 2, n=83, 85 | -46.3 (31.0) | -33.6 (42.6)
  Total Lesions, Week 4, n=83, 85 | -59.6 (30.8) | -38.5 (40.7)
  Total Lesions, Week 8, n=83, 85 | -65.7 (30.8) | -35.2 (54.0)
  Total Lesions, Week 12, n=83, 85 | -73.0 (26.7) | -47.7 (53.2)

5. Secondary Outcome: Correlation Between Skindex-29 Questionnaire Scores and Total Lesion Counts From Baseline to Week 2
Description: Analyses were performed to determine whether there was a correlation between the total lesion count and either the global or subdomain Skindex-29 questionnaire scores. Correlations between the Skindex-29 questionnaire scores and total lesion count from Baseline to Week 2 were assessed using Spearman's correlation coefficients, which ranges from -1 to 1. A score of 0 denotes no correlation, a score approaching 1 denotes correlation, and a score approaching -1 denotes inverse correlation.
Time Frame: Baseline (Week 0) and Week 2
Population: ITT Population. Missing values were imputed using the LOCF method. One participant in the Differin group had no data available and was thus excluded from analysis.
Measure: Number; unit: Correlation coefficient
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 84
Correlation coefficient
  Functional Domain | 0.042 | -0.094
  Symptomatic Domain | 0.166 | 0.002
  Emotional Domain | 0.237 | -0.137
  Global Score | 0.223 | -0.087

6. Secondary Outcome: Mean Scores for Global Change in Acne Improvement at Weeks 1, 2, 4, 8, and 12 Compared to the Start of Treatment (Prior to Week 1)
Description: Global change in acne improvement was assessed by the investigator on a 7-point scale: 1=greatly worsened, 2=significantly worsened, 3=slightly worsened, 4=no change, 5=slightly improved, 6=significantly improved, or 7=greatly improved. Global change at the indicated week was assessed in terms of change from the previous week. Change at Week 2, for example, was an assessment of change from Week 1.
Time Frame: Start of treatment and Weeks 1, 2, 4, 8, and 12
Population: ITT Population. Missing values were imputed using the LOCF method. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 82 | 84
scores on a scale
  Week 1, n=82, 82 | 5.2 (1.0) | 4.9 (0.9)
  Week 2, n=82, 83 | 5.4 (1.0) | 5.3 (0.9)
  Week 4, n=82, 83 | 5.7 (1.2) | 5.3 (1.1)
  Week 8, n=82, 83 | 5.8 (1.3) | 5.1 (1.4)
  Week 12, n=82, 84 | 6.0 (1.2) | 5.5 (1.3)

7. Secondary Outcome: Mean Scores for Self-evaluation of Acne Improvement at Weeks 1, 2, 4, 8, and 12 Compared to the Start of Treatment (Prior to Week 1)
Description: Participants self-evaluated their acne improvement on a 3-point scale: 1=worsened, 2=no changes, and 3=improved.
Time Frame: Start of treatment and Weeks 1, 2, 4, 8, and 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 82 | 84
scores on a scale
  Week 1, n=82, 82 | 2.8 (0.5) | 2.5 (0.7)
  Week 2, n=82, 83 | 2.8 (0.5) | 2.7 (0.6)
  Week 4, n=82, 83 | 2.7 (0.6) | 2.7 (0.6)
  Week 8, n=82, 83 | 2.8 (0.5) | 2.5 (0.7)
  Week 12, n=82, 84 | 2.8 (0.5) | 2.6 (0.7)

8. Secondary Outcome: Mean Acne Grades at Baseline and Weeks 1, 2, 4, 8, and 12 Assessed by the Leeds Revised Acne Grading System
Description: The acne grade on the participant's face was assessed by the investigator using the LRAG, a photographic scale allowing for the assessment of the clinical status for acne severity for the face, back, and chest. It consists of a 12-grade scale (1, least severe; 12, most severe) for inflammatory visible lesions (les.). For non-inflammatory les., this scale comprises 3 photos of les. of increasing severity (grades 1-3). The scale provides a qualitative assessment of superficial/visible les. and provides consistency and inter-/intra-rater reliability. Grading was performed prior to les. counting.
Time Frame: Baseline (Week 0); Weeks 1, 2, 4, 8, and 12
Population: ITT Population. Missing values were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 85
scores on a scale
  Baseline (Week 0) | 2.7 (0.9) | 2.6 (0.8)
  Week 1 | 2.4 (0.9) | 2.3 (0.8)
  Week 2 | 2.0 (0.8) | 2.1 (0.9)
  Week 4 | 1.7 (0.9) | 1.9 (0.8)
  Week 8 | 1.6 (0.9) | 1.9 (0.9)
  Week 12 | 1.2 (0.9) | 1.6 (1.0)

9. Secondary Outcome: Mean Change From Baseline to Weeks 1, 2, 4, 8, and 12 in Tolerance Symptoms of Peeling, Erythema, and Dryness
Description: Tolerance symptoms of peeling (flaking), erythema (redness of skin), and dryness were evaluated at each visit by the investigator. Possible scores were: 0=absent, 1=mild intermittent, 2=mild persistent, 3=moderate intermittent, 4=moderate persistent, 5=severe intermittent, and 6=severe persistent.
Time Frame: Baseline (Week 0); Weeks 1, 2, 4, 8, and 12
Population: ITT Population. Missing values were imputed using the LOCF method (i.e., the last available observation was used to estimate subsequent missing data points).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 85
scores on a scale
  Peeling, Week 1 | 0.5 (0.8) | 0.8 (1.0)
  Peeling, Week 2 | 0.2 (0.5) | 0.6 (1.1)
  Peeling, Week 4 | 0.3 (0.6) | 0.6 (1.0)
  Peeling, Week 8 | 0.1 (0.4) | 0.5 (0.9)
  Peeling, Week 12 | 0.1 (0.3) | 0.4 (0.8)
  Erythema, Week 1 | 0.6 (1.0) | 0.8 (1.1)
  Erythema, Week 2 | 0.3 (0.8) | 0.9 (1.2)
  Erythema, Week 4 | 0.3 (0.6) | 0.7 (1.0)
  Erythema, Week 8 | 0.3 (0.6) | 0.6 (1.0)
  Erythema, Week 12 | 0.2 (0.5) | 0.4 (0.9)
  Dryness, Week 1 | 0.6 (1.1) | 0.8 (1.0)
  Dryness, Week 2 | 0.4 (0.8) | 0.8 (1.2)
  Dryness, Week 4 | 0.3 (0.6) | 0.7 (1.0)
  Dryness, Week 8 | 0.2 (0.5) | 0.6 (1.1)
  Dryness, Week 12 | 0.1 (0.4) | 0.4 (0.9)

10. Secondary Outcome: Mean Change From Baseline to Weeks 1, 2, 4, 8, and 12 in Tolerance Symptoms of Itching and Burning
Description: Tolerance symptoms of itching and burning were evaluated at each visit by participants. Possible scores were: 0=absent, 1=mild intermittent, 2=mild persistent, 3=moderate intermittent, 4=moderate persistent, 5=severe intermittent, and 6=severe persistent.
Time Frame: Baseline (Week 0); Weeks 1, 2, 4, 8, and 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 83 | 85
scores on a scale
  Itching, Week 1 | 0.4 (0.8) | 0.9 (1.3)
  Itching, Week 2 | 0.2 (0.6) | 0.7 (1.0)
  Itching, Week 4 | 0.2 (0.5) | 0.7 (1.2)
  Itching, Week 8 | 0.1 (0.4) | 0.6 (1.2)
  Itching, Week 12 | 0.1 (0.3) | 0.5 (1.1)
  Burning, Week 1 | 0.3 (0.7) | 0.9 (1.3)
  Burning, Week 2 | 0.1 (0.4) | 0.6 (1.1)
  Burning, Week 4 | 0.1 (0.4) | 0.5 (1.2)
  Burning, Week 8 | 0.1 (0.2) | 0.6 (1.2)
  Burning, Week 12 | 0.0 (0.2) | 0.5 (1.1)

11. Secondary Outcome: Number of Participants in the Indicated Categories for Overall Tolerance at Week 12/Early Termination
Description: Participants were evaluated for overall tolerance to study drug by the investigator at the end of the study (Week 12 or Early Termination). Participants were given the tolerance grades of poor, fair, good, or excellent.
Time Frame: Week 12 or Early Termination
Population: ITT Population. Some participants had no data available and were thus excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Duac Gel | Differin Gel
Number analyzed (Participants) | 80 | 83
participants
  Poor | 0 | 5
  Fair | 4 | 14
  Good | 42 | 47
  Excellent | 34 | 17

ADVERSE EVENTS:
Arm/Group | Duac Gel | Differin Gel
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/85
Other Adverse Events (participants affected / at risk) | 13/83 | 22/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duac Gel (N=83) | Differin Gel (N=85)
Application Site Erythema (General disorders) | 2 | 5
Application Site Exfoliation (General disorders) | 2 | 4
Application Site Pruritus (General disorders) | 2 | 4
Application Site Dryness (General disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 0
Application Site Irritation (General disorders) | 0 | 5
Application Site Eczema (General disorders) | 0 | 4
Application Site Dermatitis (General disorders) | 0 | 2
Application Site Pain (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Puncture Site Infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.